CLINICAL TRIAL: NCT03493477
Title: Evaluation of Gingival Biotypes and Width of Keratinized Gingiva of Anterior Teeth in Adults With Abnormal Skeletal Jaw Relations: A Cross-sectional Study
Brief Title: Evaluation of Gingival Biotypes of Anterior Teeth in Adults With Abnormal Skeletal Jaw Relations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed magdy Mohamed Sabrah, Principal Investigator, Cairo University
Other Study IDs: CEBD-CU-2018-03-20
Record Dates: First submitted 2018-03-20; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Abnormal Jaw Relations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Skeletal Class II Group: From the lateral cephalometric radiograph , Steiner analysis (ANB angle should be higher than mean value, mean value 3 ±2), Witt's appraisal should be higher than mean value (mean value zero), and McNamara analysis (A-B diff NV should be higher than mean value, mean value 4±2).At least two of the three mentioned analyses should verify skeletal class II relation
  Interventions: Other: exposure will be abnormal skeletal jaw relations
- Skeletal Class III Group: From the lateral cephalometric radiograph , Steiner analysis (ANB angle should be lower than mean value, mean value 3 ±2), Witt's appraisal should be lower than mean value (mean value zero), and McNamara analysis (A-B diff NV should be lower than mean value, mean value 4±2).At least two of the three mentioned analyses should verify skeletal class III relation
  Interventions: Other: exposure will be abnormal skeletal jaw relations

INTERVENTIONS:
Other: exposure will be abnormal skeletal jaw relations — Class II skeletal jaw relation or class III skeletal jaw relation based on lateral cephalometric radiograph

SUMMARY:
The aim of this study is to evaluate gingival biotypes and width of keratinized gingiva in the anterior region of adults with abnormal skeletal jaw relations.

DETAILED DESCRIPTION:
This study will include consecutive adult patients seeking orthodontic treatment with skeletal Class II and Class III jaw relations based on clinical and cephalometric values. Each group will be further divided according to their vertical skeletal pattern. Gingival biotype will be determined -using the probe transparency method- into either thick or thin biotype for all anterior teeth in both jaws. Width of keratinized gingiva will be measured from the muco-gingival junction to the free gingival margin in the middle of the crown of the maxillary and mandibular anterior teeth using a digital caliper with a sensitivity of 0.01 mm. Statistical analysis will be applied to see the correlation between gingival biotypes , width of keratinized gingiva , and abnormal skeletal jaw relations.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients having an age range of 18 -30 years.
2. Adults with skeletal Class II and Class III jaw relation
3. Fair oral hygiene with absence of any active periodontal disease.
4. Patients with full permanent dentition (with the exception of third molars) with acceptable alignment of teeth.
5. Absence of systemic disease (medically free patients).

Exclusion Criteria:

1. Patients with extensive restorations on the anterior teeth.
2. Subjects taking medication affecting the periodontal tissues
3. History of previous periodontal surgery or orthodontic treatment.
4. Pregnant or lactating female patients
5. Syndromic patients

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Patients attending the orthodontic clinic in the orthodontic department, Faculty of Dentistry, Cairo University , who have either skeletal class II or class III maxillo-mandibular jaw relations
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between gingival biotypes and abnormal sagittal skeletal jaw relations. | 6 months
  Gingival biotype will be determined using the probe transparency method, in which probing is done in the sulcus at the mid facial aspect of maxillary and mandibular incisors and canines by a periodontal probe. Gingival thickness will be classified as thin when the underlying periodontal probe outline can be seen through the gingiva; otherwise, it will be considered thick. Results of the twelve anterior teeth will be recorded for each patient in a tabulated form. Statistical Analysis will be done to detect the correlation between gingival biotypes (Thick or thin ) and abnormal sagittal skeletal jaw relation ( skeletal class II or skeletal class III 9

SECONDARY OUTCOMES:
Correlation between width of keratinized gingiva in the anterior region and abnormal sagittal skeletal jaw relation | 6 months
  Width of keratinized gingiva will be measured from the muco-gingival junction to the free gingival margin in the middle of the crown of the maxillary and mandibular anterior teeth using a digital caliper with a sensitivity of 0.01 mm. Statistical analysis will be done to detect the correlation between the width of keratinized gingiva and abnormal sagittal jaw relations (skeletal class II or skeletal class III )
Correlation between gingival biotypes and abnormal vertical skeletal jaw relations. | 6 months
  will be determined using the probe transparency method, in which probing is done in the sulcus at the mid facial aspect of maxillary and mandibular incisors and canines by a periodontal probe. Gingival thickness will be classified as thin when the underlying periodontal probe outline can be seen through the gingiva; otherwise, it will be considered thick. Results of the twelve anterior teeth will be recorded for each patient in a tabulated form.Statistical analysis will be done to detect the correlation between the gingival biotype ( thick or thin ) and abnormal vertical skeletal jaw relations ( long face or short face )
Correlation between width of keratinized gingiva and abnormal vertical skeletal jaw relations. | 6 months
  Width of keratinized gingiva will be measured from the muco-gingival junction to the free gingival margin in the middle of the crown of the maxillary and mandibular anterior teeth using a digital caliper with a sensitivity of 0.01 mm .Statistical analysis will be done to detect the correlation between the width of keratinized gingiva and abnormal vertical skeletal jaw relations ( long face or short face )

IPD SHARING:
Plan to Share IPD: Yes